CLINICAL TRIAL: NCT00291044
Title: HSV Seroprevalence and Diagnosis of Genital Herpes in Pregnant Women
Status: Completed | Type: Observational
Sponsor: Stony Brook University (Other)
Other Study IDs: VAL R116
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Pregnancy
Keywords: pregnancy, genital herpes
MeSH Terms: conditions — Herpes Genitalis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective

INTERVENTIONS:
Other: testing for HSV 1 and 2 IgG type specific antibosy

SUMMARY:
Brief summary: The current management guidelines recommended by ACOG rely on history as a screening method to determine pregnant women who are at risk for transmitting herpes to their newborn. History fails completely in identifying the women most at risk of transmitting herpes to their newborn - the seronegative woman who acquires a primary infection from her partner during pregnancy. Despite recent advances, both pregnant women and newborns continue to be at risk of acquiring herpes infection. Genital herpes infections are epidemic in the United States. In the early 1990's, 25% of women in the US were seropositive for the HSV-2 antibody. These numbers are likely higher now. The incidence of neonatal herpes in the US cannot be accurately estimated since it is not a reportable disease. However, in some areas of the US, the incidence is 1 in 3,200 live births which would translate to an incidence of approximately three infants a day in the US . In other areas of the US, the incidence is even higher, approaching 1 in 1,500 liveborns. This protocol examines patient acceptance of HSV-1 and HSV-2 type specific serologic testing and assesses patient counseling tools. In addition, seroprevalence of HSV-2 in pregnant patients will be collected and evaluated.

DETAILED DESCRIPTION:
Detailed Description: Despite recent advances, both pregnant women and newborns continue to be at risk of acquiring herpes infection. Genital herpes infections are epidemic in the United States. In the early 1990's, 25% of women in the US were seropositive for the HSV-2 antibody (Fleming, 1997). These numbers are likely higher now. The incidence of neonatal herpes in the US cannot be accurately estimated since it is not a reportable disease. However, in some areas of the US, the incidence is 1 in 3,200 live births which would translate to an incidence of approximately three infants a day in the US (Brown, 2003). In other areas of the US, the incidence is even higher, approaching 1 in 1,500 liveborns (Whitley, personal communication, December 2002).

The current management guidelines recommended by ACOG (Guidelines for Perinatal Care, 2002) rely on history as a screening method to determine pregnant women who are at risk for transmitting herpes to their newborn. Based on data reported in NHANES III, history is an unreliable method of determining those who are infected with genital herpes (Fleming, 1997). Most importantly, history fails completely in identifying the women most at risk of transmitting herpes to their newborn - the seronegative woman who acquires a primary infection from her partner during pregnancy.

Since at-risk women can now be accurately identified by new and more accurate type-specific serologic tests, effective prevention strategies should be instituted to minimize risk of transmission to the neonate. The first obligation is to diagnose who is at risk. The highest risk is that of neonatal transmission from a mother experiencing a primary genital HSV-1 or HSV-2 infection in late pregnancy. Studies indicate that approximately 1.3% of women seroconvert during pregnancy and, among those who do, the risk of neonatal transmission is as high as 30 - 50% (Brown 1991). Conversely, the rate of neonatal transmission from women with recurrent genital herpes infection is low (<1%) (Brown, 1991, 1997; Smith, 1998; Arvin, 1986; Fonnest, 1997). However, since genital herpes is so common, the total number of cases of neonatal herpes from women with recurrent disease remains high (Fleming, 1997; STD Guidelines, 2002). Once a mother is identified as being infected with HSV-2, the health care providers - both pediatrician and obstetrician - can be alerted to the potential risk of neonatal herpes.

Management of pregnant women with or without herpes infections should include steps designed to minimize the risk of herpes transmission to neonates. This protocol examines patient acceptance of HSV-1 and HSV-2 type specific serologic testing and assesses patient counseling tools. In addition, seroprevalence of HSV-2 in pregnant patients will be collected and evaluated.

STUDY DESIGN

This is a non-treatment study of acceptance rates of HSV-1 and HSV-2 type specific serologic testing by pregnant women and their partners. This study will also evaluate Health Care Provider time spent in counseling, effectiveness of counseling tools/sessions, and acceptance of antiviral suppression by pregnant women and/or their partners. In addition, HSV-2 seroprevalence will be assessed. This study will be conducted at a single center (Obstetrics and Gynecology Office) and is not designed to yield nationally representative estimates of HSV-2 seroprevalence rates.

Pregnant women who present for their first prenatal visit will be invited to enroll. A total of 300 patients will be enrolled.

The clinician or staff will describe the study to the patient based on the provided description.

If the patient is interested in participating in the study, she will be given an informed consent to sign, told that the blood test is to determine whether she is seropositive or seronegative for genital herpes (HSV-2) and the virus that causes cold sores (HSV-1), and given a demographic form to complete. If the patient is willing to be tested for HSV-1 and HSV-2, she will continue with counseling and completion of questionnaires. For those patients willing to be tested, counseling and questionnaires will be completed during visit 1 and visit 2. For those patients who are unwilling to be tested, counseling and questionnaires will be administered during this first visit.

The investigator and office staff will monitor time spent in each counseling session, and also provide assessment of effectiveness and satisfaction with counseling tools.

STUDY ASSESSMENTS AND PROCEDURES

Screening and Assessments

Prior to inviting the patient to take part in the clinical trial, each patient's chart should be reviewed to be certain that the patient does not have a known history of genital herpes or prior knowledge of HSV-2 seropositivity.

Prior to enrollment of patients in the study, the investigator and appropriate study personnel will be provided with training on HSV serologic testing and provided with the counseling tools. This will ensure that all patients receive standardized HSV counseling at the initial visit and during the follow-up visit when test results are discussed.

It is important to note that ideally, the same person on staff should administer the Counseling Scripts using verbiage consistent with the provided scripts This should be administered with care and concern in a private setting. The counselor then should give the patient sufficient time to ask questions.

Following is an outline of study assessments and procedures Visit #1

* The clinician or staff will describe the study to the patient by the following script:

This study involves your willingness to have a blood test to determine if you are infected with the virus that causes genital herpes or the virus that causes cold sores. If you decide to participate in this study and decide to have the blood test or even if you decide NOT to have the blood test, you will be asked to complete questionnaires and counseling sessions given by the office staff. This will be a time commitment of about 1 hour and may include an additional 20 minute office visit next week.

* All patients willing to be a part of the study will sign an informed consent
* Patients will complete a Demographics Questionnaire

Patients willing to be tested will:

* Sign informed consent for blood test
* Have blood drawn for serological assessment via the FOCUS HerpeSelect 1 and 2 ELISA assay.
* Receive counseling
* Complete Questionnaire on Understanding Counseling
* Age, race and infection history will be documented on the CRF based on information from the patient's chart and the medical history sheet routinely used by the clinic (completed by the patient)
* Be given brochure and one-page information sheet
* Instruct the patient to read the entire brochure but to also focus on Page 4, the section related to pregnancy
* Schedule visit in one week (Visit 2)

Patients unwilling to be tested will:

* Complete Questionnaire about Barriers to Testing
* Receive counseling
* After receipt of counseling the patient will be asked again if willing to be tested
* If willing to be tested o Go to list of "patients willing to be tested, sign the informed consent for the blood test and draw the blood test without further counseling at this visit.
* If not willing to be tested

  o Complete Understanding of Counseling and Survey on Satisfaction with Counseling

  o Be given brochure and one-page information sheet

  o Instruct the patient to read the entire brochure but to also focus on Page 4, the section related to pregnancy

  o Repeat barriers questionnaire

  o Schedule next visit (continue with prenatal visits consistent with standard of care)
  * At next visit, ask again if willing to be tested (if yes, clinic staff will proceed with assessments and procedures under patients willing to be tested [above] except third bullet point, Receive Counseling and sixth bullet point Complete questionnaire Understanding Counseling. Offer the patient the brochure and information sheet again.
  * If at any point during the study the patient changes her mind and becomes willing to be tested, document the reason for this change in the CRF.
* Investigator/staff will document time spent for counseling in the case report form

Follow Up Assessment

Visit #2

Patients willing to be tested will:

* Be given results of the HSV-1 and HSV-2 serologic test
* Receive Counseling

  1. Patients with negative HSV-2 serologic test If the woman is HSV-1 seronegative, counsel her with the section of the Script: For patients who are HSV-1 seronegative
* Encourage the patient to discuss her test results and its meaning with her partner
* Ask the following question (answer will be documented in the case report form by Yes/No response):

  * Do you know if your partner is positive for HSV-1 or HSV-2 . If NO to either HSV-1 and HSV-2, follow up as described below.

Follow-up visit

• During normally scheduled pre-natal visits (up to week 28), ask the patient if her partner had been tested. Document answer in the case report form.

OR

2. Patients with positive HSV-2 serologic test If the woman is HSV-1 seronegative, counsel her with the section of the Script: For patients who are HSV-1 seronegative

* Encourage the patient to discuss her test results and its meaning with her partner

  o Give the patient the brochure (Taking Charge of your Life and instruct the patient to read the entire brochure but to also focus on the section related to pregnancy
* Ask the following questions (answer will be documented in the case report form by Yes/No response):

  * Are you willing to take medicine to treat your herpes during your pregnancy?
  * Do you know if your partner is positive for HSV-1 or HSV-2 . If NO to either HSV-1 or HSV-2, follow up as described below.

Follow-up visit

* During normally scheduled prenatal visits (up to week 28), ask the patient if her partner had been tested. Document answer in the case report form.
* Complete Understanding Counseling Questionnaire [appropriate questionnaire for seronegative or seropositive patients, respectively] and Survey of Satisfaction with Counseling,

Investigator/counseling staff will:

• Document time spent for counseling and for ordering HSV-1 and HSV-2 blood tests for each patient in the case report form Upon completion of study, complete Satisfaction with Counseling Tools Questionnaire

HEALTH OUTCOMES

At the first visit a self administered questionnaire regarding barriers to testing will be given to each eligible patient refusing to be tested. After counseling, this questionnaire will be repeated for those patients who still refuse testing. All patients will be counseled and will be given two self administered questionnaires. One questionnaire will assess the patient's understanding of the counseling and the other will assess the patient's satisfaction with the counseling session. At the second visit, those patients who were tested will receive their test results and will be counseled on their status (positive or negative). These patients will receive two self administered questionnaires. One questionnaire will assess the patient's understanding of counseling (specific to their status), and the other will assess the patient's satisfaction with the counseling session. A separate self administered questionnaire will be given to the investigator and/or appropriate office personnel to assess their satisfaction with the counseling tools and sessions.

DATA ANALYSIS AND STATISTICAL CONSIDERATIONS

Hypotheses

This is a non-treatment study in pregnant women to assess the acceptances of HSV serologic testing and their understanding and satisfaction with counseling tools.

Interim Analysis

An interim analysis is not planned.

Primary Analysis

• The percentage of pregnant patients who accept HSV-1 and HSV-2 type specific testing

Secondary Analyzes

* The mean (SD) percent and frequencies (n, %) of questions answered correctly by all subjects in the "Understanding Counseling" questionnaire
* The mean (SD) percent and frequencies (n, %) of questions answered correctly by seronegative subjects in the "Understanding Counseling" questionnaire
* The frequencies (n, %) and mean (SD) percent of questions answered correctly by seropositive subjects in the "Understanding Counseling" questionnaire
* The frequencies (n, %) and mean (SD) scores for each item in the "Satisfaction with Counseling" (for the patient) scale
* The frequencies (n, %) and mean (SD) scores for each item in the "Satisfaction with Counseling Tools" ( for the counselor) scale
* The percentage of partners of pregnant women who were tested
* The percentage of pregnant women (who are HSV-2 positive) who would accept antiviral suppressive therapy during pregnancy
* The frequencies (n, %) and mean (SD) scores for each reason/item in the "Reason For Choosing Not To Be Tested" scale
* The mean (SD) total time (in minutes) spent by the investigator and clinic staff in obtaining the both the HSV-2 type specific serologic test and counseling

ELIGIBILITY:
Inclusion Criteria:

* pregnant 24 weeks or less

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant subjects
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2005-09; Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
% of patients willing to be tested

SECONDARY OUTCOMES:
Barriers to be tested for HSV

CONTACTS AND LOCATIONS:
Overall Officials: David A Baker, MD, Principal Investigator — Stony Brook University
Locations (1):
- Dept ObGyn, 6 Tech Dr, Stony Brook, New York, United States

REFERENCES:
- [Background] Arvin AM, Hensleigh PA, Prober CG, et al. Failure of antepartum maternal cultures to predict the infant's risk of exposure to herpes simplex virus at delivery. N Engl J Med 1986; 315:796-800. 2. Brown ZA, Benedetti J, Ashley R, et al. Neonatal herpes simplex virus infection in relation to asymptomatic maternal infection at the time of labor. N Engl J Med 1991; 324:1247-1252. 3. Brown ZA, Selke S, Zeh J, et al. The acquisition of herpes simplex virus during pregnancy. N Engl J Med 1997; 337:509-515. 4. Brown ZA, Wald A, Morrow RA, et al. Effect of Serologic Status and Cesarean Delivery on Transmission Rates of Herpes Simplex Virus from Mother to Infant. JAMA 2003; 289:203-209. 5. Fleming DT, McQuillan GM, Johnson RE, et al. Herpes simplex virus type 2 in the United States, 1976 to 1994. N Engl J Med 1997; 337:1105-1111. 6. Fonnest G, de la Fuente Fonnest I, Weber T. Neonatal herpes in Denmark 1977-1991. Acta Obstet Gynecol Scand 1997; 76:355-358. 7. Guidelines for Perinatal Care: AAP, ACOG, 2002. pp. 292-297. 8. Sexually Transmitted Disease Treatment Guidelines 2002. MMWR 2002; 51:12- 9. Smith JR, Cowan FM, Munday P. The management of herpes simplex virus infection in pregnancy. Br J Obstet Gynaecol 1998; 105:255-260.